CLINICAL TRIAL: NCT06761495
Title: Is Isthmosel Becoming History? The Effect of Three Different Uterotomy Closure
Brief Title: Can Cesarean Scar Defects be Prevented?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MLP Tokat
Record Dates: First submitted 2024-12-19; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Isthmocele
Keywords: niche; baseball suturing; uterotomy; caesarean section

STUDY DESIGN:
Intervention Model Description: Caesarean section patients were eligible for the study and randomized preoperatively into 3 different uterotomy closure techniques (baseball, single-locked and single-unlocked groups). In all 3 groups, No. 1 absorbable multiflament polyglactin 910(Vicryl, Ethicon Inc, Somerville, NJ, USA) suture thread was used to close the uterine incision. When necessary, haemostatic additional sutures were applied using the same material.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isthmosel (caesarean scar defect ) (Active Comparator): Isthmosel or caesarean scar defect is a poch-like defect in the myometrium at the isthmic level that is thought that it might occur as a result of insufficient healing process of the uterine incision after caesarean section.
  Interventions: Procedure: Baseball Suturing Technique; Procedure: Single-Layer Locked Continuous Suturing Technique; Procedure: Single-Layer Unlocked Continuous Suturing Technique
- Residual myometrial thickness (Active Comparator): Three months after the operation, residual myometrial thickness localization was evaluated by ultrasonography.
  Interventions: Procedure: Baseball Suturing Technique; Procedure: Single-Layer Locked Continuous Suturing Technique; Procedure: Single-Layer Unlocked Continuous Suturing Technique

INTERVENTIONS:
Procedure: Baseball Suturing Technique — (Baseball Suturing Technique): A corner suture was placed at the right corner of the incision. Next, the second stitch was placed at the apex of the left corner and tied with a knot. Then, the free end of the suture was cut and running baseball stitch pattern was started. The suturing pattern was performed by taking bites from the inside out through the upper and lower lips of the wound at approximately 1 cm intervals with a 1 cm margin from the wound edges
Procedure: Single-Layer Locked Continuous Suturing Technique — (Single-Layer Locked Continuous Suturing Technique): A corner suture was placed at the right corner of the incision. Next, the second stitch was placed at the apex of the left corner and tied with a knot. Then, the free end of the suture was cut and single-layer-locked continuous suturing was started. The suturing pattern was performed by taking bites from outside to inside through the lower lip and inside to outside through the upper lip of the wound. Each time, a lock was formed by passing through the loop formed by the previous suture. The suturing was performed at approximately 1 cm intervals with a 1 cm margin from the wound edges
Procedure: Single-Layer Unlocked Continuous Suturing Technique — (Single-Layer Unlocked Continuous Suturing Technique): The uterotomy line was closed in a single-layer continuous suturing pattern that is explained above as group 2 but without passing the needle through the loop formed by the previous sutu

SUMMARY:
In this study, uterotomy after cesarean section was performed using 3 different suture techniques and aimed to demonstrate the potential of the baseball suture technique to prevent the isthmusel complication known as cesarean scar defect.

DETAILED DESCRIPTION:
An isthmocoele or cesarean scar defect is a pit-like defect in the myometrium at the isthmic level, thought to be the result of inadequate healing of the uterine incision after cesarean section. It is important not to underestimate isthmocele and to take preventive measures as it can lead to serious gynecologic and obstetric complications. However, which suturing technique is best in preventing isthmocele formation has not yet been established. The aim of this study was to compare the effects of 3 different uterine closure techniques on isthmocele formation during cesarean section.

In this study, a total of 120 term (>37 weeks) pregnant women with no previous cesarean section and scheduled for primary cesarean section will be randomized preoperatively to 3 different uterotomy closure techniques (baseball, single-lock and non-single-lock groups).

ELIGIBILITY:
Inclusion criteria:

* Pregnant women undergoing C/S for the first time
* 37 weeks < gestation (term pregnancies)

Exclusion Criteria:

* Presence of regular contractions in the uterus
* Cervical dilatation of more than 4 cm, indicating the onset of the active phase of labour
* Placental abnormalities
* Previous uterine surgery
* Multiple pregnancy
* Premature rupture of membranes
* Chorioamnionitis
* Preoperative haemoglobin level below 10g/dl
* Body mass index (BMI) above 35kg/m2
* Any comorbidity (e.g. diabetes, hypertension, pre-eclampsia, eclampsia)
* Smoking and/or alcohol use
* The need for a blood transfusion.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 120 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Isthmocele was be evaluated | Three months postoperatively
  The presence and anatomical location of isthmocele were be evaluated by ultrasonography.

CONTACTS AND LOCATIONS:
Overall Officials: Neset Gumusburun, M.D., Principal Investigator — Gazıosmanpasa Unıversity
Locations (1):
- Gazıosmanpasa Unıversity, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF
Time Frame: The data that support the findings of this study are available on request from corresponding author.